CLINICAL TRIAL: NCT07169006
Title: The Effect of Preoperative Gabapentin on Postoperative Pain Control and Analgesic Requirements Following Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: MD326/2024
Record Dates: First submitted 2025-09-05; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-01

CONDITIONS: Bariatric Surgery Analgesia

STUDY DESIGN:
Intervention Model Description: Assuming an effect size of 0.5 for preoperative gabapentin, a sample of 51 patients in each group would be enough to detect such effect, if true, at 0.05 alpha error and 0.80 power of the test
Who Masked: Participant
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 (Experimental): Will receive a single dose of gabapentin 300 mg preoperatively before standard general anesthesia
  Interventions: Drug: Group 1
- Group 2 (Placebo Comparator): will receive a placebo before standard general anesthesia
  Interventions: Drug: Group 2

INTERVENTIONS:
Drug: Group 1 — Will receive a single dose of gabapentin 300 mg preoperatively before standard general anesthesia
  Other Names: Gabapentin 300
  Arms: Group 1
Drug: Group 2 — will receive a placebo before standard general anesthesia
  Other Names: Placebo
  Arms: Group 2

SUMMARY:
The importance of bariatric anesthesia and analgesia research cannot be ignored as it can inform and improve the perioperative protocols for other patients with morbid obesity irrespective of the surgical procedures they are undergoing

DETAILED DESCRIPTION:
Among various postoperative complications, pain is the main adverse event experienced by patients. Good control of postoperative pain is an important factor for reducing early postoperative complications such as pulmonary embolism, deep vein thrombosis, ileus, and respiratory infections, and for decreasing length of stay, lowering costs, and increasing patient satisfaction

ELIGIBILITY:
Inclusion criteria:

* patients with American Society of Anesthesiologists physical status ASA I to III
* both genders
* Morbid obese scheduled for bariatric surgery

Exclusion Criteria:

* patients with impaired liver or kidney disease
* patients with history of hypersensitivity to gabapentin
* patients with history of alcohol abuse, chronic pain or frequent use of analgesic
* patients with uncontrolled medical disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 102 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Comparing pain score between the two groups during 1st postoperative 24 hours using visual analogue score (VAS | 24 hours postoperative
  Comparing pain score between the two groups during 1st postoperative 24 hours using visual analogue score (VAS